CLINICAL TRIAL: NCT02857153
Title: Comparsion of the Effect of High Versus Low Mean Arterial Pressure (MAP) Levels on Clinical Outcomes in Elderly Patients During Noncardiothoracic Surgery Under General Anesthesia
Brief Title: Effect of High vs. Low MAP Levels on Clinical Outcomes in Elderly Patients During Noncardiothoracic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hu Anmin (Other)
Collaborators: West China Hospital (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Taihe Hospital (Other); The Third Affiliated Hospital of Kunming Medical College. (Other); Sichuan Provincial People's Hospital (Other); Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Hu Anmin, Shenzhen People's Hospital, The Second Clinical Medical College of Jinan University
Organization: The Second Clinical Medical College of Jinan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016001
Record Dates: First submitted 2016-07-15; First posted 2016-08-05 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Aging; Surgery; Blood Pressure; Anesthesia; Blood Loss, Surgical; Postoperative Delirium
Keywords: MAP; Blood loss; Postoperative delirium; Elderly patients; Noncardiothoracic surgery
MeSH Terms: conditions — Blood Loss, Surgical; Emergence Delirium; Hemorrhage | interventions — urapidil; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-level MAP (Experimental): According to grouping, MAP is regulated to the goal level (60-70 mmHg) during general anesthesia.
  Interventions: Drug: Urapidil; Drug: Phenylephrine; Procedure: Low-level MAP
- High-level MAP (Experimental): According to grouping, MAP is regulated to the goal level (90-100 mmHg) during general anesthesia.
  Interventions: Drug: Urapidil; Drug: Phenylephrine; Procedure: High-level MAP

INTERVENTIONS:
Drug: Urapidil — If necessary, intravenous urapidil 0.2-0.5 mg/kg when mean arterial pressure exceeded 10 mmHg of the target value, rather than more anesthesia, may be used in situations wherein sympathetic stimulation was high; yet a sufficient amount of anesthesia was being administered and bispectral index showed an adequate depth of hypnosis. Sedation was provided by a propofol infusion targeted to a BIS number of approximately 50 during general anesthesia.
  Other Names: Ebrantil
Drug: Phenylephrine — If necessary, intravenous phenylephrine 4-6 μg/kg when mean arterial pressure exceeded 10 mmHg of the target value, rather than more anesthesia, may be used in situations wherein sympathetic stimulation was high; yet a sufficient amount of anesthesia was being administered and bispectral index showed an adequate depth of hypnosis. Sedation was provided by a propofol infusion targeted to a BIS number of approximately 50 during general anesthesia.
  Other Names: Metaoxedrin; Neosynephrine
Procedure: Low-level MAP — MAP is regulated to the goal level (60-70 mmHg) during general anesthesia.
  Arms: Low-level MAP
Procedure: High-level MAP — MAP is regulated to the goal level (90-100 mmHg) during general anesthesia.
  Arms: High-level MAP

SUMMARY:
This will be a multicentre, randomised, controlled and prospective clinical trial. All participants provided their written informed consent to participate in a randomized trial that examined the effects of low-level MAP (60-70 mmHg) vs. high-level MAP (90-100 mmHg) in elderly patients (65 or more years of age) during noncardiothoracic surgery under general anesthesia. The investigators hypothesise high-level blood presure of the intervention for reducing the incidence of post-operative complications.

DETAILED DESCRIPTION:
This will be a multicentre, randomised, controlled and prospective clinical trial. Elderly patients will be included from seven centers, including Shenzhen People's Hospital affiliated to Jinan University, West China Hospital affiliated to Sichuan University, Taihe Hospital affiliated to Hubei University of Medicine, The Third Affiliated Hospital of Kunming Medical University, Sichuan Provincial People's Hospital, Guizhou Provincial People's Hospital and Henan Provincial People's Hospital. This research protocol was approved by the Institutional Review Board of Jinan University (2016001).

On the day of surgery, patients come to the operating room and are provided with standard monitoring. General anesthesia is given using midazolam and propofol, opioids, muscle relaxants and maintained with sevoflurane with inhaled concentrations of 1.5% sevoflurane in oxygen. Supplemental dosing of 1 μg/kg of fentanyl is used every hour from induction up to approximately 1 hour prior to the end of surgery. A tramadol bolus of 2 mg/kg is given 15 to 30 mins before the end of surgery. Propofol infusion is stopped 5 to 10 mins prior to the end of surgery, whereas at the end of skin closure, remifentanil was discontinued.

According to grouping, MAP is regulated to the goal level (60-70 mmHg or 95-100 mmHg) during general anesthesia. If necessary, intravenous antihypertensives (urapidil or phenylephrine when mean arterial pressure exceeded 10 mmHg of the target value), rather than more anesthesia, may be used in situations wherein sympathetic stimulation was high; yet a sufficient amount of anesthesia was being administered and bispectral index showed an adequate depth of hypnosis. Sedation was provided by a propofol infusion targeted to a BIS number of approximately 50 during general anesthesia. Atropine and esmolol would be used at the time of heart rate <50 beats/min and >110 beats/min, respectively.

Lactated Ringer's solution was given to bring the maintenance fluids to 10 ml/kg/h. Blood loss could be corrected for in a 1:1 ratio using gelofusine. Hospital transfusion guidelines were used to determine whether blood products were necessary (haemoglobin level less than 10 g/dl in patients with cardiac comorbidities, and below 7 g.dl-1 in those without cardiac disease). For later starting cases, an additional bolus of Ringer's solution of 1.5 ml/kg/fasted hour from 8 AM was given to bring the total 2 ml/kg/fasted hour. If urine output decreased to <0.5 mL/kg/h for 1 hour, fursemide 0.3 mg/kg was given.

Mechanical ventilation patterns are adjusted to obtain an end-tidal carbon dioxide value of 35-45 mmHg, at 5-10 min after induction of anesthesia.

For patients with endotracheal tubes, intravenous sedatives including propofol or midazolam were administrated continuously and titrated by bedside nurses to a target sedation level. Daily awakening is used for those who were not extubated in the morning.

All patients receive patient controlled intravenous analgesia during postoperative days 1 to 3.

ELIGIBILITY:
Inclusion Criteria:

* male and females, American Society of Anesthesiologists I-II-III, 65 or more years of age, scheduled to undergo noncardiothoracic surgery with general anesthesia are enrolled.

Exclusion Criteria:

* the patient suffered from Cardiovascular Disease and Metabolic Diseases, such as hypertension, cardiac disease, diabetes;
* the patient has severe liver, kidney or blood disease;
* the patient is accompanied severe cognitive impairment (Mini-Mental State Examination (MMSE) score < 15);
* preoperative history of schizophrenia, epilepsy, parkinsonism, use of cholinesterase inhibitor, or levodopa treatment;
* use of haloperidol or other neuroleptics during or after anesthesia;
* neurosurgery;
* individuals unlikely to survive for >24 hrs; previous participation in this study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 322 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of delirium | Within the first 7 days after surgery

SECONDARY OUTCOMES:
Delirium duration days (Postoperative delirium defined by the confusion assessment method for the ICU (CAM-ICU)) | Within the first 7 days after surgery
Intra-operative blood loss | Intra-operative
  Estimate of blood loss occurring during the surgical procedure as determined by anesthesia staff and documented by anesthesia, nursing and surgical staff as per hospital protocol.
Intraoperative urine volume. | Intra-operative
All-cause 28-day mortality. | The investigators would observe it within the 28-day period after surgery.
  Outcome assessment will be performed by independent researchers.

CONTACTS AND LOCATIONS:
Overall Officials: Hu Anmin, Study Director — Jinan University
Locations (7):
- China (7):
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Taihe Hospital affiliated to Hubei University of Medicine, Shiyan, Hubei
  - West China Hospital affiliated to Sichuan University, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The Third Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] London MJ. Intraoperative Mean Blood Pressure and Outcome: Is 80 (mmHg) the "New" 60? Anesthesiology. 2016 Jan;124(1):4-6. doi: 10.1097/ALN.0000000000000923. No abstract available. PMID 26540150
- [Result] Monk TG, Bronsert MR, Henderson WG, Mangione MP, Sum-Ping ST, Bentt DR, Nguyen JD, Richman JS, Meguid RA, Hammermeister KE. Association between Intraoperative Hypotension and Hypertension and 30-day Postoperative Mortality in Noncardiac Surgery. Anesthesiology. 2015 Aug;123(2):307-19. doi: 10.1097/ALN.0000000000000756. PMID 26083768
- [Result] Walsh M, Devereaux PJ, Garg AX, Kurz A, Turan A, Rodseth RN, Cywinski J, Thabane L, Sessler DI. Relationship between intraoperative mean arterial pressure and clinical outcomes after noncardiac surgery: toward an empirical definition of hypotension. Anesthesiology. 2013 Sep;119(3):507-15. doi: 10.1097/ALN.0b013e3182a10e26. PMID 23835589
- [Result] Chang HS, Hongo K, Nakagawa H. Adverse effects of limited hypotensive anesthesia on the outcome of patients with subarachnoid hemorrhage. J Neurosurg. 2000 Jun;92(6):971-5. doi: 10.3171/jns.2000.92.6.0971. PMID 10839257
- [Result] Reich DL, Bennett-Guerrero E, Bodian CA, Hossain S, Winfree W, Krol M. Intraoperative tachycardia and hypertension are independently associated with adverse outcome in noncardiac surgery of long duration. Anesth Analg. 2002 Aug;95(2):273-7, table of contents. doi: 10.1097/00000539-200208000-00003. PMID 12145033
- [Derived] Hu A, Qiu Y, Zhang P, Hu B, Yang Y, Li S, Zhao R, Zhang Z, Zhang Y, Zheng Z, Qiu C, Li F, Gong X. Comparison of the effect of high versus low mean arterial pressure levels on clinical outcomes and complications in elderly patients during non-cardiothoracic surgery under general anesthesia: study protocol for a randomized controlled trial. Trials. 2017 Nov 21;18(1):554. doi: 10.1186/s13063-017-2233-8. PMID 29162132